CLINICAL TRIAL: NCT06528132
Title: Social Worker-led Mindfulness-based Intervention for Managing Depressive Symptoms in Community-dwelling Older Adults in Hong Kong: A Randomised Controlled Trial
Brief Title: Social Worker-led Mindfulness-based Intervention for Older People
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); Christian Family Service Centre (Other); The Mental Health Association of Hong Kong (Other); The Salvation Army, Hong Kong and Macau Command (Other); Haven of Hope Hospital (Other); Hong Kong Sheng Kung Hui (Unknown); Tung Wah Group of Hospitals (Other); Aberdeen Kai-fong Welfare Association (Other); Hong Kong Society for the Aged (Unknown); Neighbourhood Advice-Action Council (Other)
Responsible Party: Principal Investigator, Professor Terry Y.S. Lum, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA220105A
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Depressive Symptoms
Keywords: Modified mindfulness-based intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants in the intervention group will receive mindfulness-based intervention from social workers either with or without peer supporters involved. The care as usual group will receive usual service provided in District Elderly Community Centres (DECC) and Integrated Community Centre for Mental Wellness (ICCMW).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- social worker-led MBI (enhanced with peer supporters) (Experimental): Participants in the social worker-led modified MBI group will receive mindfulness training from social workers. In addition, they will receive support from peer supporters.
  Interventions: Behavioral: Mindfulness-based intervention (MBI) (enhanced with peer supporters)
- social worker-led MBI (without peer supporters) (Experimental): Participants in the social-worker led modified MBI group will receive mindfulness training from social workers.
  Interventions: Behavioral: Experimental: social worker-led MBI (without peer supporters)
- Care as usual group (No Intervention): The care as usual group will receive usual service provided in District Elderly Community Centres (DECC) and Integrated Community Centre for Mental Wellness (ICCMW).

INTERVENTIONS:
Behavioral: Mindfulness-based intervention (MBI) (enhanced with peer supporters) — Mindfulness-based intervention combines mindfulness meditation with cognitive behavioural therapy (CBT) elements to reduce or prevent recurrent major depressive disorders. On-site support and regular follow-up by peer supporters.
  Arms: social worker-led MBI (enhanced with peer supporters)
Behavioral: Experimental: social worker-led MBI (without peer supporters) — Mindfulness-based intervention combines mindfulness meditation with cognitive behavioural therapy (CBT) elements to reduce or prevent recurrent major depressive disorders.
  Arms: social worker-led MBI (without peer supporters)

SUMMARY:
Preliminary findings from a previous study conducted by the investigators suggest that a task-shared approach with modified mindfulness-based cognitive therapy (MBCT) supported by social workers is beneficial in managing depressive symptoms and improving mindful non-reactivity among older adults. However, the possibility for social workers to lead a mindfulness-based intervention (MBI) independently to improve its scalability and service accessibility remains unclear. The project aims to:

1. Evaluate the effectiveness of social worker-led MBI in improving depression in older adults with mild to moderate depressive symptoms as compared to care as usual;
2. Examine the effectiveness of incorporating peer supporters in social worker-led MBI compared to those without peer supporters;
3. To identify potential mechanisms of change in MBI for depressive symptoms.

DETAILED DESCRIPTION:
Mindfulness-based cognitive therapy (MBCT) is a promising approach to managing a series of health and psychological conditions among older adults. To increase its acceptability, feasibility, and scalability, MBCT has been adapted and delivered in a variety of formats. Apart from delivering the intervention in person by a certified mindfulness teacher, MBCT has been adapted to be self-taught, delivered online, or partially led by social workers.

In a previous study conducted by the investigators, it was found that a task-shared approach with modified MBCT supported by social workers is effective in producing change in older adults' mental health and mindfulness. However, whether social workers are competent to lead a mindfulness-based intervention (MBI) informed by MBCT on their own and produce effective changes in outcome measures pertaining to mental health remains unclear.

Furthermore, the effects of incorporating peer supporters into mental health interventions are unclear. The uses and implementation of peer support across mental health contexts vary greatly and the effects are mixed. In a pilot study on men with advanced prostate cancer, it has been suggested that the presence of peer support in modified mindfulness-based cognitive therapy group intervention may reinforce intervention effects. Furthermore, in an online intervention for older adults with elevated depressive symptoms, peer support has been found to improve engagement and adherence to the intervention. However, in a systematic review and meta-analysis, it has been found that while incorporating one-to-one peer support in mental health services has a modest positive impact on self-reported psychosocial outcomes such as self-rated recovery and empowerment, there is no evidence for improvement in clinical outcomes.

With the growing older people population and a need for greater social welfare capacity to promote older adults' well-being, the current study aims to examine the effectiveness of social worker-led MBI informed by MBCT in improving depression in older adults with mild to moderate depressive symptoms. In addition, the effectiveness of incorporating peer supporters into the intervention will be examined.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* have depressive symptoms of mild level or above, as indicated by scoring 5-14 on PHQ-9
* can give informed consent to participate

Exclusion Criteria:

* known history of autism, intellectual disability, schizophrenia-spectrum disorder, bipolar disorder, Parkinson's disease, or dementia
* current abuse of drugs or alcohol
* difficulty in communication
* imminent suicidal risk
* timing or training is unsuitable for the participant

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2026-03-16 (Estimated)

PRIMARY OUTCOMES:
Change from baseline depression at Week 6 and Week 18 | Baseline and Week 6, Week 18
  Depression will be measured by the validated Chinese version of the Patient Health Questionnaire (PHQ-9). The total score will be used, ranging from 0 to 27. Higher scores indicate higher levels of depressive symptoms.
Change from baseline anxiety at Week 6 and Week 18 | Baseline and Week 6, Week 18
  Anxiety will be measured by the validated Chinese version of the Generalized Anxiety Disorder scale (GAD-7). The total score will be used, ranging from 0 to 21. Higher scores indicate higher levels of anxiety symptoms.

OTHER OUTCOMES:
Change from baseline mindfulness at Week 6 and Week 18 | Baseline and Week 6, Week 18
  Mindfulness will be measured by the Chinese validated Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF). The total score of the FFMQ-SF (ranging from 20 to 100) as well as the sum (ranging from 4 to 20) of the five subscales (i.e., observe, describe, acting with awareness, nonjudging, and nonreactivity) will be used. Higher scores indicate higher mindfulness.
Change from baseline stress at Week 8 and Week 18 | Baseline and Week 6, Week 18
  Stress will be measured by a single-item subjective level of stress (SLS-1), which is rated on a scale from 0 to 10. A higher score indicates a greater subjective level of stress
Change from baseline quality of life at Week 6 and Week 18 | Baseline and Week 6, Week 18
  Health-related quality of life will be measured by the European Quality of life 5 Dimensions 5 Level Version (EQ-5D-5L) in traditional Chinese. The measure assesses five dimensions of health (i.e., mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) at five levels (no problem, slight problems, moderate problems, severe problems, and extreme problems). An index value ranging from 0 to 1 will be used, with a score closer to 1 indicating a better health state. Current self-rated health will be measured using a visual analogue scale ranging from 0 to 100, with higher scores indicating better self-rated health.
Change from baseline self-compassion at Week 6 and Week 18 | Baseline and Week 6, Week 18
  Self-compassion will be measured by the Chinese version of the Self-Compassion Scale-Short Form (SCS-SF). The total score will be used, ranging from 12 to 60. Higher scores indicate higher self-compassion.
Change from baseline rumination at Week 6 and Week 18 | Baseline and Week 6, Week 18
  Rumination will be measured by the Brooding Subscale of the Ruminative Response Scale (RRS-10 Chinese version). The total score will be used, ranging from 5 to 20. Higher scores indicate a greater rumination tendency.
Change from baseline self-efficacy at Week 6 and Week 18 | Baseline and Week 6, Week 18
  Self-efficacy will be measured by the Chinese version of the General Self-Efficacy Scale. The total score will be used, ranging from 10 to 40. Higher scores indicate greater self-efficacy.
Change from baseline resilience at Week 6 and Week 18 | Baseline and Week 6, Week 18
  Resilience will be measured by the Chinese version of the 2-item Connor-Davidson Resilience Scale (CD-RISC2). The total score will be used, ranging from 0 to 8. Higher scores indicate higher resilience.
Change from baseline general health status at Week 6 and Week 18 | Baseline and Week 6, Week 18
  General health status will be assessed using one non-comparative and two comparative questions pertaining to health. Health status will be measured on a scale ranging from 0 to 4. Higher scores indicate poorer health status.

CONTACTS AND LOCATIONS:
Overall Officials: Terry YS Lum, PhD, Principal Investigator — Department of Social Work and Social Administration, The University of Hong Kong
Locations (13):
- Hong Kong (13):
  - Hong Kong Society for the Aged, Eastern District
  - HKSKH Lok Man Alice Kwok Integrated Service Centre, Kowloon City
  - SKH Holy Carpenter Church, Kowloon City
  - The Mental Health Association of Hong Kong, Kwun Tong
  - Haven of Hope District Elderly Community Service, Sai Kung
  - Wellness Zone - Integrated Community Centre for Mental Wellness, Sai Kung
  - HKSKH Western District Elderly Community Centre, Sai Wan
  - TWGHs Lok Hong Integrated Community Centre for Mental Wellness, Sai Wan
  - Wilson T.S. Ｗang District Elderly Community Centre, Shatin
  - Aberdeen Kai-fong Welfare Association, Southern District
  - The Salvation Army Taipo Multi-Service Centre for Senior Citizens, Tai Po
  - The Neighbourhood Advice-Action Council, Tuenmen
  - SKH Wong Tai Sin District Elderly Community Centre, Wong Tai Sin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dragomanovich HM, Dhruva A, Ekman E, Schoenbeck KL, Kubo A, Van Blarigan EL, Borno HT, Esquivel M, Chee B, Campanella M, Philip EJ, Rettger JP, Rosenthal B, Van Loon K, Venook AP, Boscardin C, Moran P, Hecht FM, Atreya CE. Being Present 2.0: Online Mindfulness-Based Program for Metastatic Gastrointestinal Cancer Patients and Caregivers. Glob Adv Health Med. 2021 Nov 3;10:21649561211044693. doi: 10.1177/21649561211044693. eCollection 2021. PMID 35174001
- [Background] Hazlett-Stevens H, Singer J, Chong A. Mindfulness-Based Stress Reduction and Mindfulness-Based Cognitive Therapy with Older Adults: A Qualitative Review of Randomized Controlled Outcome Research. Clin Gerontol. 2019 Jul-Sep;42(4):347-358. doi: 10.1080/07317115.2018.1518282. Epub 2018 Sep 11. PMID 30204557
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Lei X, Zhong M, Liu Y, Xi C, Ling Y, Zhu X, Yao S, Yi J. Psychometric properties of the 10-item ruminative response scale in Chinese university students. BMC Psychiatry. 2017 Apr 28;17(1):152. doi: 10.1186/s12888-017-1318-y. PMID 28454569
- [Background] Meng R, Yu Y, Chai S, Luo X, Gong B, Liu B, Hu Y, Luo Y, Yu C. Examining psychometric properties and measurement invariance of a Chinese version of the Self-Compassion Scale - Short Form (SCS-SF) in nursing students and medical workers. Psychol Res Behav Manag. 2019 Aug 30;12:793-809. doi: 10.2147/PRBM.S216411. eCollection 2019. PMID 31565007
- [Background] Montero-Marin J, Taylor L, Crane C, Greenberg MT, Ford TJ, Williams JMG, Garcia-Campayo J, Sonley A, Lord L, Dalgleish T, Blakemore SJ; MYRIAD team; Kuyken W. Teachers "Finding Peace in a Frantic World": An Experimental Study of Self-Taught and Instructor-Led Mindfulness Program Formats on Acceptability, Effectiveness, and Mechanisms. J Educ Psychol. 2021 Nov;113(8):1689-1708. doi: 10.1037/edu0000542. Epub 2021 Oct 18. PMID 34912129
- [Background] Ni MY, Li TK, Yu NX, Pang H, Chan BH, Leung GM, Stewart SM. Normative data and psychometric properties of the Connor-Davidson Resilience Scale (CD-RISC) and the abbreviated version (CD-RISC2) among the general population in Hong Kong. Qual Life Res. 2016 Jan;25(1):111-6. doi: 10.1007/s11136-015-1072-x. Epub 2015 Jul 22. PMID 26198665
- [Background] Smit D, Miguel C, Vrijsen JN, Groeneweg B, Spijker J, Cuijpers P. The effectiveness of peer support for individuals with mental illness: systematic review and meta-analysis. Psychol Med. 2023 Aug;53(11):5332-5341. doi: 10.1017/S0033291722002422. Epub 2022 Sep 6. PMID 36066104
- [Background] Tomasino KN, Lattie EG, Ho J, Palac HL, Kaiser SM, Mohr DC. Harnessing Peer Support in an Online Intervention for Older Adults with Depression. Am J Geriatr Psychiatry. 2017 Oct;25(10):1109-1119. doi: 10.1016/j.jagp.2017.04.015. Epub 2017 May 3. PMID 28571785
- [Background] Tong X, An D, McGonigal A, Park SP, Zhou D. Validation of the Generalized Anxiety Disorder-7 (GAD-7) among Chinese people with epilepsy. Epilepsy Res. 2016 Feb;120:31-6. doi: 10.1016/j.eplepsyres.2015.11.019. Epub 2015 Nov 28. PMID 26709880
- [Background] Wang W, Bian Q, Zhao Y, Li X, Wang W, Du J, Zhang G, Zhou Q, Zhao M. Reliability and validity of the Chinese version of the Patient Health Questionnaire (PHQ-9) in the general population. Gen Hosp Psychiatry. 2014 Sep-Oct;36(5):539-44. doi: 10.1016/j.genhosppsych.2014.05.021. Epub 2014 Jun 6. PMID 25023953
- [Background] Wang YH, Wang YL, Leung DKY, Ng ZLY, Chan OLH, Wong SMY, Chan RCL, Liu T, Wong GHY, Lum TYS. Effectiveness of an age-modified mindfulness-based cognitive therapy (MBCT) in improving mental health in older people with depressive symptoms: a non-randomised controlled trial. BMC Complement Med Ther. 2025 Feb 26;25(1):81. doi: 10.1186/s12906-025-04781-6. PMID 40011881
- [Background] Wong, S. M. Y., Lam, B. Y. H., Wong, C. S. M., Lee, H. P. Y., Wong, G. H. Y., Lui, S. S. Y., Chan, K. T., Wong, M. T. H., Chan, S. K. W., Chang, W. C., Lee, E. H. M., Suen, Y. N., Hui, C. L. M., & Chen, E. Y. H. (2021). Measuring subjective stress among young people in Hong Kong: Validation and predictive utility of the single-item subjective level of stress (SLS-1) in epidemiological and longitudinal community samples. Epidemiology and Psychiatric Sciences, 30, e61. https://doi.org/10.1017/S2045796021000445
- [Background] Zhang, J. X., & Schwarzer, R. (1995). Measuring optimistic self-beliefs: A Chinese adaptation of the General Self-Efficacy Scale. Psychologia: An International Journal of Psychology in the Orient, 38(3), 174-181.
- [Background] DeSalvo KB, Bloser N, Reynolds K, He J, Muntner P. Mortality prediction with a single general self-rated health question. A meta-analysis. J Gen Intern Med. 2006 Mar;21(3):267-75. doi: 10.1111/j.1525-1497.2005.00291.x. Epub 2005 Dec 7. PMID 16336622
- [Background] Li ZB, Lam TH, Ho SY, Chan WM, Ho KS, Li MP, Leung GM, Fielding R. Age- versus time-comparative self-rated health in Hong Kong Chinese older adults. Int J Geriatr Psychiatry. 2006 Aug;21(8):729-39. doi: 10.1002/gps.1553. PMID 16858746
- [Background] Crane PhD C, Ganguli PhD P, Ball MSc S, Taylor PhD L, Blakemore PhD SJ, Byford PhD S, Dalgleish PhD T, Ford PhD T, Greenberg PhD M, Kuyken PhD W, Lord Ma L, Montero-Marin PhD J, Sonley MEd A, Ukoumunne PhD OC, Williams PhD JMG. Training School Teachers to Deliver a Mindfulness Program: Exploring Scalability, Acceptability, Effectiveness, and Cost-effectiveness. Glob Adv Health Med. 2020 Dec 15;9:2164956120964738. doi: 10.1177/2164956120964738. eCollection 2020. PMID 33403157
- [Background] Hou J, Wong SY, Lo HH, Mak WW, Ma HS. Validation of a Chinese version of the Five Facet Mindfulness Questionnaire in Hong Kong and development of a short form. Assessment. 2014 Jun;21(3):363-71. doi: 10.1177/1073191113485121. Epub 2013 Apr 16. PMID 23596271
- [Derived] Wang YL, Wang YH, Leung DKY, Wong SMY, Ng ZLY, Chan RCL, Chan OLH, Chan WC, Wong GHY, Lum TYS. Peer-supported mindfulness-based intervention for managing depressive symptoms in community-dwelling older adults: Protocol for a randomized controlled trial. Contemp Clin Trials. 2025 Aug;155:107991. doi: 10.1016/j.cct.2025.107991. Epub 2025 Jun 20. PMID 40544956

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT06528132/Prot_SAP_001.pdf